CLINICAL TRIAL: NCT04319627
Title: Statins for Venous Event Reduction in Patients With Venous Thromboembolism
Acronym: SAVER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Eastern Norway Health Authorities RHF (Unknown); Southern health region, Norway (Unknown); Programme hospitalier de recherche clinique, France (Unknown); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAVER Trial
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism; Blood Clot; Post Thrombotic Syndrome
Keywords: Rosuvastatin; Statin; PTS; VTE
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis; Postthrombotic Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rosuvastatin (Experimental): Participants randomized to the experimental arm will take one rosuvastatin 20 mg tablet by mouth every day for the duration of their participation in the study.
  Interventions: Drug: Rosuvastatin Calcium
- Placebo (Placebo Comparator): Participants randomized to the control arm will take one placebo tablet by mouth every day for the duration of their participation in the study.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Rosuvastatin Calcium — Each participant will receive the usual treatment for their newly diagnosed blood clot in addition to the intervention they are randomized to.
  Other Names: Rosuvastatin
  Arms: Rosuvastatin
Drug: Placebo Oral Tablet — Each participant will receive the usual treatment for their newly diagnosed blood clot in addition to the intervention they are randomized to.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The standard or usual treatment for patients diagnosed with deep vein thrombosis or pulmonary embolism is treatment with blood thinners (called anticoagulants).

While treatment of blood clots with blood thinners is effective, some research has shown that adding a statin (medication used to lower cholesterol) may give extra protection. It is thought that statins can improve how cells along the walls of the vein control inflammation, which can prevent new blood clots from forming.

The medication in this study, rosuvastatin, is approved in Canada for use as a cholesterol-lowering medication. The use of rosuvastatin in this study is considered investigational. This means that Health Canada has not approved the use of rosuvastatin as a treatment for blood clots. However, it has been approved for use in this research study.

The purpose of this study is to examine if adding a statin (rosuvastatin) to the usual blood thinner treatment will decrease the risk of another blood clot forming. The investigators also hope to discover if taking a statin reduces damage to your veins. To do this, some of the participants in this study will get rosuvastatin and others will receive a placebo (a substance that looks like the study rosuvastatin but does not have any active or medicinal ingredients). The placebo in this study is not intended to have any effect on your blood clot. A placebo is used to make the results of the study more reliable.

DETAILED DESCRIPTION:
Recent research has demonstrated that it is plausible that statins have additive, and potentially even synergistic effects, in reducing recurrent VTE in patients managed with anticoagulant-based strategies. Furthermore, it is plausible that statins may reduce the risk of recurrent VTE in those not on anticoagulants and therefore offer an alternative in patients with contraindications to anticoagulants (e.g. after major intracranial bleed), who refuse to take anticoagulants long-term (e.g. due to lifestyle modifications or fear of bleeding) or who cannot afford anticoagulants (e.g. vulnerable or impoverished populations). Finally, statins may also provide protection from recurrent VTE in patients who are not fully compliant with anticoagulant therapy. However, no known RCTs have been done to explore these possibilities.

This study aims to determine if generic rosuvastatin reduces the risk of recurrent VTE compared to placebo in patients with symptomatic major VTE.

Primary Objectives

- To determine the primary outcome event rate (i.e. symptomatic recurrent major VTE [proximal DVT or segmental or larger PE]) in patients taking generic rosuvastatin compared to placebo.

Secondary Objectives

* To determine the major bleeding event rate in patients taking generic rosuvastatin compared to placebo.
* To explore if rosuvastatin reduces the incidence of PTS, as measured by the Villalta scale at end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic objectively confirmed proximal leg DVT (above the trifurcation of the popliteal vein) and/or PE (segmental or greater) diagnosed in the last 30 days.

Exclusion criteria

1. Unable or unwilling to provide written informed consent;
2. < 18 years of age;
3. Women of childbearing potential unwilling to use appropriate contraception;
4. Currently prescribed a statin;
5. A known medical history or current diagnosis of any of the following for which statins are indicated in secondary prevention:

   1. Diabetes;
   2. Abdominal aortic aneurysm;
   3. Peripheral arterial disease;
   4. Stroke;
   5. Transient ischemic attack (TIA);
   6. Myocardial infarction (MI);
   7. Acute coronary syndromes;
   8. Stable/unstable angina;
   9. Coronary or other arterial revascularization;
6. Known diagnosis of hypercholesterolemia or dyslipidemia;
7. Contraindication to rosuvastatin;

   1. Known hypersensitivity or intolerance to statins;
   2. History of muscle disorders or statin-related muscle pain;
   3. Known liver disease (active liver disease, e.g. Hepatitis A, B, C, non-alcoholic fatty liver);
   4. Chronic kidney disease (creatinine clearance < 30ml/min);
   5. Currently pregnant or breast feeding;
   6. Taking cyclosporine;
   7. Taking atazanavir/ritonavir;
   8. Taking darolutamide;
   9. Taking regorafenib;
8. Unstable medical or psychological condition that would interfere with trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Recurrent Major VTE | Up to 60 months
  Symptomatic recurrent major VTE (proximal DVT or segmental or larger PE) occurring between randomization and the end of follow-up (i.e. completion of the trial) in patients taking generic rosuvastatin as compared with placebo.

SECONDARY OUTCOMES:
Post Thrombotic Syndrome | Up to 60 months
  Post-thrombotic syndrome as measured by the Villalta scale throughout the follow-up period in patients taking generic rosuvastatin as compared with placebo. The Villalta PTS scale has been adopted by the International Society on Thrombosis and Haemostasis (ISTH) as a standard to diagnose and grade the severity of PTS in clinical studies.
  Points are summed to yield total score: 0-4: No PTS; 5-9: Mild PTS; 10-14: Moderate PTS; 15 or more, or presence of ulcer: Severe PTS.
Number of participants diagnosed with non-major VTE during follow-up | Up to 60 months
  Symptomatic non-major VTE (see below) occurring between randomization and the end of follow-up (i.e. completion of the trial) in patients taking generic rosuvastatin as compared with placebo.
  Non-major VTE:
  * Distal DVT (distal to the trifurcation of the popliteal vein);
  * Isolated sub-segmental PE;
  * Upper extremity DVT;
  * Superficial phlebitis > 5 cm;
  * Superficial phlebitis ≤ 5 cm.
Number of participants diagnosed with an arterial vascular event during follow-up | Up to 60 months
  Components of composite arterial vascular events (see below) occurring between randomization and the end of follow-up (i.e. completion of the trial) in patients taking generic rosuvastatin as compared with placebo.
  Components of composite arterial vascular events:
  * Fatal myocardial infarction;
  * Non-fatal myocardial infarction;
  * Hospitalization for unstable angina;
  * Coronary artery revascularization;
  * Sudden cardiac death;
  * Ischemic stroke.
Number of deaths during study participation | Up to 60 months
  All-cause mortality occurring between randomization and the end of follow-up (i.e. completion of the trial) in patients taking generic rosuvastatin as compared with placebo.

OTHER OUTCOMES:
Number of participants who have a bleeding event during follow-up | Up to 60 months
  Bleeding event (major, clinically relevant non-major, minor) occurring between randomization and the end of follow-up (i.e. completion of the trial) in patients taking generic rosuvastatin as compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Delluc, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (31):
- Canada (14):
  - Foothills Medical Centre, Calgary, Alberta
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - Niagara Health - St. Catharines Site, St. Catharines, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill Univeristy Health Centre, Montreal, Quebec
  - CIUSSS de-l'Ouest-de-l'Ile-de-Montreal -St. Mary's Hospital Center, Montreal, Quebec
  - CHU de Quebec-Université Laval, Québec, Quebec
- France (8):
  - CHU d'Angers - Service d'accueil et traitement des Urgences, Angers
  - Brest University Hospital Centre, Brest
  - CHU de Clermont-Ferrand, Hôpital Gabriel Montpied, Clermont-Ferrand
  - APHP Hôpital Louis Mourier, Colombes
  - CHU de Dijon - Service d'imagerie diagnostique et thérapeutique, Dijon
  - GH La Rochelle - Ré-Aunis - Service de Médecine vasculaire, La Rochelle
  - Centre Hospitalier Universitaire De Saint Etienne, Saint-Etienne
  - CHI Toulon - La Seyne sur Mer - Hôpital Sainte Musse, Toulon
- Mater Misericordiae University Hospital, Dublin, Ireland
- University of Insubria, Varese, Italy
- Ostfold Hopsital, Sarpsborg, Norway
- United Kingdom (6):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - Glasgow Royal Infirmary, Glasgow
  - King's College Hospital NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No